CLINICAL TRIAL: NCT06180369
Title: Evaluation of Clinical Efficacies of Different Agents in Molar-Incisor Hypomineralization-Affected Molars
Brief Title: Clinical Efficacies of Different Agents in Molar-Incisor Hypomineralization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MarmaraPedo3
Record Dates: First submitted 2023-12-01; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Molar-Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC Fuji Triage ® GC America Inc., Alsip, Illinois ) (Other): Fissure sealant application with GC Fuji Triage (GC America Inc., Alsip, Illinois )
  Interventions: Other: GC Fuji Triage ® GC America Inc., Alsip, Illinois )
- BeutiSealant (Shofu, Kyoto, Japonya) (Other): Fissure sealant application with BeutiSealant (Shofu, Kyoto, Japonya)
  Interventions: Other: BeutiSealant (Shofu, Kyoto, Japonya)

INTERVENTIONS:
Other: GC Fuji Triage ® GC America Inc., Alsip, Illinois ) — Fissur Sealent application
  Arms: GC Fuji Triage ® GC America Inc., Alsip, Illinois )
Other: BeutiSealant (Shofu, Kyoto, Japonya) — Fissur Sealent application
  Arms: BeutiSealant (Shofu, Kyoto, Japonya)

SUMMARY:
This study aims to assess the clinical effectiveness of GC Fuji Triage ® (GC America Inc., Alsip, Illinois) and BeutiSealant (Shofu, Kyoto, Japan) in children aged 8-13 with multiple molars affected by Molar-Incisor Hypomineralization (MIH). The comparison focuses on permanent first molars affected by MIH.

DETAILED DESCRIPTION:
The study targets children within the specified age range with MIH-affected molars, comparing the clinical outcomes of GC Fuji Triage and BeutiSealant. The assessment will provide valuable insights into the efficacy of these agents in managing severe hypomineralization, contributing to our understanding of effective treatment modalities for MIH.

The evaluation criteria include restoration success, prevention of further decay development, prevention of post-eruption breakdown, alleviation of tooth sensitivity, and measurement of life quality. These criteria will be compared with those of Resin Fissure Sealant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 8-13 with hypomineralization in their first permanent molars.
* Children without systemic diseases or developmental dental anomalies that could affect hypomineralization.
* Those with at least two molars exhibiting molar-incisor hypomineralization (MIH), specifically scoring 1 and 3 according to the MIH-Tll index.
* Children with a positive or 'definitely positive' cooperation according to the Frankl Behavior Rating Scale (Frankl et al., 1962).
* Absence of spontaneous pain, abscess, mobility, or inter-radicular lesions in the tooth to be treated.
* Patients or their parents consenting to participate in the treatment.

Exclusion Criteria:

* Children with systemic diseases or developmental dental anomalies that could affect hypomineralization.
* To have MIH outside the specified scores.
* Children unable to continue treatment in the chair due to cooperation problems.
* Failure to attend control sessions or a desire not to continue with the study.
* Patients and their parents unwilling to participate in the treatment.
* If the patient cannot attend control sessions or disrupts sessions, they will be withdrawn from the study.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The Schiff Cold Air Sensitivity Score | 1.5 -2 year
  The Schiff Cold Air Sensitivity Score is a test conducted in dental units. Cold air from a spray is applied to the surface of the tooth's dentin, 2-3 mm away, and at a 90-degree angle, with continuous pressure of 45-60 PSI for 2-3 seconds, following the isolation of neighboring teeth. The temperature should be around 20 degrees Celsius. The patient's pain level is then scored by the dentist using a scale.
  * Score 0: No response to the stimulus.
  * Score 1: Responds to the stimulus but does not request it to be stopped.
  * Score 2: Responds to the stimulus, requests it to be stopped, or makes movements to avoid it.
  * Score 3: Responds to the stimulus, finds it painful, and requests it to be stopped.
Parent Satisfaction | 1.5-2 year
  Parent Satisfaction: To assess parental satisfaction regarding the applied restoration, a Likert-type scale will be used to score crowns based on their appearance, color, shape, size, and overall aesthetic (Suguna and Gurunathan, 2021).
  1. Not satisfied at all
  2. Not satisfied
  3. Neither satisfied nor dissatisfied (Neutral)
  4. Satisfied
  5. Very satisfied